CLINICAL TRIAL: NCT00613067
Title: The Amplitude Change of the Auditory Evoked N1 Component as a Predictor of Response to Escitalopram Treatment in Patients With Generalized Anxiety Disorder
Brief Title: ERP N1 as a Treatment Predictor of Generalized Anxiety Disorder
Acronym: N1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Seung-Hwan Lee, Department of Psychiatry, Inje Univ. Ilsanpaik Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB-0709-053
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized anxiety disorder; N100; Central serotonergic activity
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GAD (Experimental): 35 patients with Generalized Anxiety disorder
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram — * Start with escitalopram 10mg
  * According to patient's symptoms, stay on 10mg or increase up to 20mg
  * Concomitant therapy : up to Xanax 0.5mg, or Ativan 1mg, not allowed above these dosages
  * Length of washout period will be at least 2 weeks for any psychotropic drugs
  Other Names: lexapro

SUMMARY:
Amplitude changes of the N1 and the N1/P2 ERP component in response to different tone intensities have been suggested as a correlative of central serotonergic activity. A strong loudness dependence amplitude increase (strong intensity dependence) reflects low serotonergic neurotransmission and vice versa. Many researchers assumed that the brain serotonergic activity could influence treatment response of highly selective serotonin reuptake inhibitors in depression and anxiety disorders. There are a couple of studies reporting associations of N1 amplitude intensity dependence with response to Citalopram (positive correlation) and Reboxetine (negative correlation) treatment in major depressive disorder patients. But so far there have been no reports about associations between ERP N1 and antidepressant response in GAD patients.

So, it would be very interesting to explore the correlations between ERP N1 amplitude change and the Escitalopram treatment responsiveness in GAD patients.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV TR for GAD
* Hamilton Rating Scale for Anxiety (HAMA) >18
* 18 to 75 years old

Exclusion Criteria:

* Severe medical illness
* Other psychiatric illness
* HAMD > 18
* High suicidal risk
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Event related potential (ERP) N100 | Baseline

SECONDARY OUTCOMES:
- HAMA - HAMD - CGI - Beck Anxiety Inventory(self rating) | baseline, 2, 4, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hwan Lee, MD, PhD, Principal Investigator — Psychiatry department, Inje Univ. Ilsanpaik Hospital; Young-Min Park, MD, PhD, Study Director — Psychiatry department, Inje Univ. Ilsanpaik Hospital; Sung-Man Bae, PhD, Study Director — Psychiatry department, Inje Univ. Ilsanpaik Hospital
Locations (1):
- Psychiatry department, Inje Univ. Ilsanpaik Hospital, Goyang, Kyunggi, South Korea

REFERENCES:
- [Result] Linka T, Muller BW, Bender S, Sartory G, Gastpar M. The intensity dependence of auditory evoked ERP components predicts responsiveness to reboxetine treatment in major depression. Pharmacopsychiatry. 2005 May;38(3):139-43. doi: 10.1055/s-2005-864126. PMID 15902586
- [Result] Linka T, Sartory G, Bender S, Gastpar M, Muller BW. The intensity dependence of auditory ERP components in unmedicated patients with major depression and healthy controls. An analysis of group differences. J Affect Disord. 2007 Nov;103(1-3):139-45. doi: 10.1016/j.jad.2007.01.018. Epub 2007 Feb 20. PMID 17316822
- [Result] Linka T, Muller BW, Bender S, Sartory G. The intensity dependence of the auditory evoked N1 component as a predictor of response to Citalopram treatment in patients with major depression. Neurosci Lett. 2004 Sep 9;367(3):375-8. doi: 10.1016/j.neulet.2004.06.038. PMID 15337269